CLINICAL TRIAL: NCT01926236
Title: A Phase III, Randomised, Multicentre Open-label Study of Active Symptom Control (ASC) Alone or ASC With Oxaliplatin/ 5F-U Chemotherapy for Patients With Locally Advanced/ Metastatic Biliary Tract Cancers Previously Treated With Cisplatin/ Gemcitabine Chemotherapy.
Brief Title: Active Symptom Control Alone or With mFOLFOX Chemotherapy for Locally Advanced/ Metastatic Biliary Tract Cancers
Acronym: ABC06
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Principal Investigator, Juan Valle, Medical Oncologist, The Christie NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTSp048; A16281 (Other Grant/Funding Number: Cancer Research UK (CTAAC)); 2013-001812-30 (EudraCT Number)
Record Dates: First submitted 2013-08-17; First posted 2013-08-20 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Biliary Tract Cancer; Gallbladder Cancer; Cholangiocarcinoma; Ampullary Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Gallbladder Neoplasms; Cholangiocarcinoma | interventions — Leucovorin; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Active symptom control (ASC) (Active Comparator): Active Symptom Control
  Interventions: Other: Active Symptom Control
- Arm B: ASC with OxMdG chemotherapy (Experimental): Active Symptom Control with OxMdG chemo (Oxaliplatin, L-folinic acid & 5FU)
  Interventions: Other: Active Symptom Control; Drug: L-folinic acid; Drug: 5 FU; Drug: Oxaliplatin

INTERVENTIONS:
Other: Active Symptom Control — Active Symptom Control: monthly clinical review and active symptom control as needed, including biliary drainage, antibiotics, analgesia, steroids, anti-emetics, other palliative treatment for symptom control, palliative radiotherapy, blood transfusion.
Drug: L-folinic acid — L-folinic acid 175mg (or folinic acid 350mg) q14d, up to 12 cycles
  Other Names: Folinic acid
  Arms: Arm B: ASC with OxMdG chemotherapy
Drug: 5 FU — 5 FU 400 mg/m2 (bolus), 2400 mg/m2 (infusion), q 14d, up to 12 cycles
  Other Names: Fluorouracil
  Arms: Arm B: ASC with OxMdG chemotherapy
Drug: Oxaliplatin — Oxaliplatin 85mg/m2, q 14d, up to 12 cycles
  Other Names: Eloxatin
  Arms: Arm B: ASC with OxMdG chemotherapy

SUMMARY:
The purpose of this study is to determine whether fit patients (with ECOG performance score of 0-1) with advanced biliary tract cancer (ABC) benefit from chemotherapy in the second-line setting (after prior therapy with cisplatin and gemcitabine) in terms of overall survival.

DETAILED DESCRIPTION:
Active chemotherapy drugs for the treatment of ABC include gemcitabine, fluoropyrimidines and platinum agents. The randomized NCRN phase III ABC-02 trial provided level A evidence supporting first-line combination cisplatin and gemcitabine (CisGem) chemotherapy in ABC. To date, there is no randomized data to support the use of second-line chemotherapy in ABC. In this setting only a small number of retrospective and prospective (phase II) studies employing multiple different chemotherapy schedules have been conducted (level C). Thus, active symptom control (ASC) is the current standard of care after development of resistance to first-line chemotherapy. Oxaliplatin has activity in several gastrointestinal tumours and has synergistic activity with a favourable toxicity profile when used in combination with 5-FU. Several studies using mFOLFOX for biliary tract tumours have provided promising efficacy data and acceptable toxicity.

The aim of this trial is to determine if patients with ABC benefit with respect to survival from the addition of mFOLFOX chemotherapy to ASC in the second-line setting after progression to first-line treatment with CisGem. This study will establish the standard of care for patients with ABC who have progressed on first line CisGem chemotherapy.

This is a randomised phase III, multi-centre, controlled, open-label trial of patients with advanced biliary tract cancer with evidence of disease progression after prior CisGem chemotherapy treatment. Eligible patients (ECOG 0-1, adequate haematological, renal and liver function, adequate biliary drainage, with no evidence of ongoing infection) will be randomized to receive either ASC ("standard" arm) or ASC with oxaliplatin/5-FU chemotherapy ("experimental" arm). The total number of participants planned is 162 (randomized 1:1). At randomisation the following factors will be controlled for: serum albumin level, platinum sensitivity (determined from first-line therapy) and locally advanced vs metastatic disease.

The primary end point is overall survival. Quality of life and economic evaluation will assess the impact on patients and relative cost effectiveness of the intervention. Archival paraffin-embedded tissue will be collected at baseline and prospective blood samples (whole blood, serum and plasma) will be collected for translational research.

ELIGIBILITY:
Inclusion Criteria:

* Histologically / cytologically verified, non-resectable or recurrent / metastatic cholangiocarcinoma, gallbladder or ampullary carcinoma.
* Patients must have failed no more than one prior course of chemotherapy (gemcitabine and cisplatin) with clear evidence of disease progression.
* ECOG performance status 0-1.
* Age >=18 years and life expectancy >3 months.
* Adequate renal function with serum urea and serum creatinine < 1.5 times upper limit of normal (ULN) and creatinine clearance >= 30ml/min
* Adequate haematological function: Hb >= 100g/l, WBC >= 3.0 x 10*9/L, ANC >= 2 x 10*9/L, platelet count >= 100 x 10*9/L
* Adequate liver function: total bilirubin < 60 μmol/L and ALP, along with AST and/or ALT ≤ 5 x ULN
* Adequate biliary drainage, with no evidence of ongoing infection (patients on maintenance antibiotics are eligible when acute sepsis has resolved).
* Women of child bearing age must have a negative pregnancy test prior to study entry and be using an adequate contraception method, which must be continued for 4 months after the study, unless child bearing potential has been terminated by surgery/radical radiotherapy
* Men must be willing to use an adequate method of contraception during chemotherapy and until 6 months after chemotherapy
* Patients must have given written informed consent
* Patients must be randomised and those allocated chemotherapy must start treatment within 6 weeks of diagnosis of disease progression

Exclusion criteria:

* Incomplete recovery from previous therapy or unresolved biliary tree obstruction (includes ongoing neuropathy of grade >1 from cisplatin)
* Any evidence of severe or uncontrolled systemic diseases which, in the view of the investigator, makes it undesirable for the patient to participate in the trial
* Evidence of significant clinical disorder or laboratory finding which, in the opinion of the investigator makes it undesirable for the patient to participate in the trial
* Any patient with a medical or psychiatric condition that impairs their ability to give informed consent
* Any other serious uncontrolled medical conditions
* Clinical evidence of metastatic disease to brain
* Any pregnant or lactating woman
* Clinically significant cardiovascular disease. [i.e. active; or <12 months since e.g. cerebrovascular accident, myocardial infarction, unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, uncontrolled hypertension].

  **Hypertension grading of ≥ 3 is an exclusion criteria (CTCAE v4.03). However, patients who have controlled hypertension with medication and/or diet may be included at the investigator's discretion. (This should be noted in the medical history section of the CRF).
* Patients must not have a history of other malignant diseases within the last 5 years (other than adequately treated non-melanotic skin cancer or in-situ carcinoma of the uterine cervix).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2014-02; Primary Completion 2018-01-05 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | Evaluated by monthly follow-up until 12 months after last patient included

SECONDARY OUTCOMES:
Progression-free survival | Evaluated by monthly follow-up until 12 months after last patient included
  Clinical progression assessed monthly, radiological progression assessed to RECIST criteria every 12 weeks for patients in the chemotherapy arm.
Response rate (chemotherapy arm only) | After 12 weeks of treatment
Toxicity (frequency of adverse events and serious adverse events) | Evaluated monthly until 12 months after last patient included
  Events will be classified according to CTCAE V4.03
Quality of life | Evaluated every 3 months until 12 months after last patient included
  Assessed from patient completed questionnaire data: QLQ-C30 and QoL BiL
Costs of health and social care | Evaluated every 3 months until 12 months after last patient included
Health status (Euroqol) | Evaluated every 3 months until 12 months after last patient included
Quality adjusted life years (QALYs) | Evaluated every 3 months until 12 months after last patient included
  Estimated from Euroqol and survival using published utility tariffs

CONTACTS AND LOCATIONS:
Overall Officials: Juan Valle, Prof, Principal Investigator — The Christie NHS Foundation Trust
Locations (17):
- United Kingdom (17):
  - Queen Elizabeth Hospital, Birmingham
  - Bristol Haematology & Oncology Centre, Bristol
  - North Cumbria University Hospitals, Carlisle
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Castle Hill Hospital, Hull
  - St James' Hospital, Leeds
  - Clatterbridge Cancer Centre, Liverpool
  - Guy's and St Thomas' Hospital, London
  - Hammersmith Hospital, London
  - Royal Free Hospital, London
  - University College London, London
  - Maidstone Hospital, Maidstone
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Weston Park Hospital, Sheffield
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Lamarca A, Palmer DH, Wasan HS, Ross PJ, Ma YT, Arora A, Falk S, Gillmore R, Wadsley J, Patel K, Anthoney A, Maraveyas A, Iveson T, Waters JS, Hobbs C, Barber S, Ryder WD, Ramage J, Davies LM, Bridgewater JA, Valle JW; Advanced Biliary Cancer Working Group. Second-line FOLFOX chemotherapy versus active symptom control for advanced biliary tract cancer (ABC-06): a phase 3, open-label, randomised, controlled trial. Lancet Oncol. 2021 May;22(5):690-701. doi: 10.1016/S1470-2045(21)00027-9. Epub 2021 Mar 30. PMID 33798493